CLINICAL TRIAL: NCT02125110
Title: Effect of Prenatal Exposure to Neurotoxicants on the Developing Brain: an MRI Study
Brief Title: PERINE : Effect of Prenatal Exposure to Neurotoxicants on the Developing Brain : an MRI Study
Acronym: PERINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2013-A01420-45
Record Dates: First submitted 2014-04-22; First posted 2014-04-29 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Effects of Neurotoxicants on the Brain
Keywords: neurotoxicants; MRI; developing brain
MeSH Terms: interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- study group (cohort PELAGIE) (Experimental): 100 children included in the cohort PELAGIE
  Interventions: Device: MRI; Other: neuropsychological assessment
- pilot group (no cohort PELAGIE) (Experimental): 10 children not included in the PELAGIE cohort to optimise MRI
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI
Other: neuropsychological assessment
  Arms: study group (cohort PELAGIE)

SUMMARY:
This project aims at evaluating the consequences of prenatal exposure to neurotoxicants (solvents, organophosphate pesticides) on the developing brain, in children aged from 10 to 12 years.

ELIGIBILITY:
Inclusion Criteria:

* Children included in the cohort PELAGIE
* Children participated in the study PEPSY
* Age between 10 and 12 years (pilot study)

Exclusion Criteria:

* Maternal smoking and or alcohol consumption during pregnancy (study group)
* Children with a health event affecting neurodevelopment
* Children treated with methylphenidate, psychotropic or anti-epileptics

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 112 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Measurement of the brain activity and its functionality | day 1
  Measurement of the fractional anisotropy of the regions of interest on MRI :
  - with DTI (Diffusion Tensor Imaging) : DTI can be used to generate quantitative maps of the scalar (anisotropy, based on measurements of FA and mean diffusivity (MD)) or tensor (diffusivity expressed in the form of a 3x3 matrix) type. An intergroup analysis will be carried out to identify regions with FA and MD values different between exposed and non-exposed subjects. Tractography of the fibre bundles in the white matter could also be carried out, based on regions of interest extracted, for example, from high resolution morphometry or functional activation maps. The connectivity between these different regions may also be studied.

SECONDARY OUTCOMES:
Measurement of the brain activity and its functionality | day 1
  Measurement of the cerebral blood flow and the activation of the regions of interest on MRI with :
  * BOLD-fMRI (Blood Oxygen Level Dependent) : detection of the voxels activated, for each child, during the tasks (motor inhibition (Go / No-Go), attention (Posner's task) and working memory (N-back)) and comparison of levels of brain activation between exposure groups
  * ASL (Arterial Spin Labeling) : quantitative value for cerebral blood flow
Results of neuropsychological tests | day 1
  Correlation between the results of neuropsychological tests (subtests of the NEPSY (developmental NEuroPSYchological assessment) and the WISC-IV (Wechsler Intelligence Scale for Children version IV) tests that will evaluate motor inhibition, attention, working memory and graphomotor capacities) and MRI measurement

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Rennes, Rennes, France

REFERENCES:
- [Result] Binter AC, Bannier E, Simon G, Saint-Amour D, Ferre JC, Barillot C, Monfort C, Cordier S, Chevrier C, Pele F. Prenatal exposure to glycol ethers and motor inhibition function evaluated by functional MRI at the age of 10 to 12 years in the PELAGIE mother-child cohort. Environ Int. 2019 Dec;133(Pt A):105163. doi: 10.1016/j.envint.2019.105163. Epub 2019 Sep 11. PMID 31518935